CLINICAL TRIAL: NCT05926713
Title: Evaluate the Effect of Dietary Supplement Combined Supervised Exercise on Physical Performance and Body Composition Among Patients With Sarcopenia and Severe Sarcopenia Comorbid With COPD or ILD: A Prospective, Multi-center Cohort Study
Brief Title: Evaluate the Effect of Dietary Supplement Combined Exercise Among Patients With Sarcopenia Comorbid With Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OEP-Sarcojoint
Record Dates: First submitted 2022-11-22; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Sarcopenia; COPD; ILD
MeSH Terms: conditions — Sarcopenia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nutritional supplements and supervised exercise on Sarcopenia group and Severe Sarcopenia group (Experimental): The intervention consisted of providing nutritional supplements and supervised exercise for 12 weeks. After the intervention (the 12th week), the trial commissioned company provides nutritional supplements with a market price of about NT$4,000 per month for three months free to participants who are willing to continue taking the products. Those participants will be tracked for one year.
  Interventions: Dietary Supplement: Sarcojoint®; Behavioral: supervised exercise

INTERVENTIONS:
Dietary Supplement: Sarcojoint® — All participants are administered Sarcojoint® containing leucinine 1 g, arginine 1.5 g, Vitamin D 7.5μg, chondroitin 400 mg, calcium 300 mg, and glucosamine 700 mg per package, and take 1 package twice a day.
Behavioral: supervised exercise — All participants are required to walk 6500 steps every day for 12 weeks, and the data are recorded by Xiaomi-smart-band.

SUMMARY:
This trial is a prospective multi-center study. The purpose of this study is to evaluate the effect of dietary supplement combined with supervised exercised on the physical performance, body composition and lung function among patients with Sarcopenia and severe Sarcopenia in chronic lung disease. After participants enroll in this study, 12-week clinical trial will be conducted to analyze the improvement regarding Sarcopenia and different severity of Sarcopenia before and after the intervention of exercise and nutritional products, which can further provide reference for clinical intervention and rehabilitation.

DETAILED DESCRIPTION:
The design of clinical trial

This study is a prospective, multi-center, and non-invasive cohort study. All participants are diagnosed with COPD or ILD with Sarcopenia or severe Sarcopenia. The intervention consisted of providing nutritional supplements and supervised exercise for 12 weeks. After the intervention (the 12th week), the trial commissioned company provides nutritional supplements with a market price of about NT$4,000 per month for three months free to participants who are willing to continue taking the products. Those participants will be tracked for one year. The primary purpose of the study is to investigate improvement of physical performance, body composition and lung function before and after the intervention. The secondary purpose of the study is to compare the effect of the same intervention on Sarcopenia and different severity of Sarcopenia regarding the improvement of physical performance, body composition and lung function. Furthermore, the subgroup analysis is conducted to compare those who achieve the exercise requirement with those who do not concerning their physical performance, body composition and lung function.

Trail procedures

1. Baseline demographic characteristic, health behavior and exercise habits are collected by questionnaires.
2. The main disease diagnosis, medication, clinical assessment questionnaire or biochemical examination and radiological examination results are collected.
3. According to the 2019 Asian Sarcopenia Consensus, participants are examined by SARC-Calf questionnaire, grip strength test and a physical performance test, including sit-stand test, short physical performance battery (SPPB), gait speed test and six-minute walk test. Afterward, bioelectrical impedance analysis (BIA) and Dual-energy X-ray absorptiometry (DXA) are applied to all participants to analyze body composition. Participants are classified into Sarcopenia group and severe Sarcopenia group.
4. All patients receive pulmonary function test and blood test ( complete blood count, hepatic function, including [CHOL、TG、UA、SGOT、SGPT、ALK、BIL、TOTAL.BIL、DIRECT、LDH], renal function [BUN、CREAT、CA、CL、NA、K、T、P、ALB], Albumin, Vitamin D before and after the trail.
5. All participants are administered Sarcojoint® containing leucinine 1 g, arginine 1.5 g, Vitamin D 7.5μg, chondroitin 400 mg, calcium 300 mg, and glucosamine 700 mg per package, and take 1 package twice a day.
6. All participants are required to walk 6500 steps every day for 12 weeks, and the data are recorded by Xiaomi-smart-band.
7. The research nurse provides health education and a recording handbook for exercise and dietary record to participants before the intervention. During the intervention, the research nurse tracks participants' compliance and records the adverse reaction by telephone interview at the first week, and every other week.
8. At the 12th week, all participants receive a comprehensive functional assessment as that at baseline after intervention to investigate the intervention effect on different severity of Sarcopenia.
9. At the 12th week, trial commissioned manufacturer provide nutritional supplements free for 3 months. Those patients will be continuously tracked for the follow-up data for the post hoc analysis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with COPD (chronic obstructive pulmonary disease) or ILD (interstitial lung disease) from Department of Chest medicine in Taichung Veterans General Hospital, judged by the doctor that they do not need hospitalization or emergent treatment.
* Outpatients who meet the diagnostic criteria for Sarcopenia after evaluation by a physician.

Exclusion Criteria:

* Patients who refuse to sign the consent form
* Patients who are under 20 years old
* Patients who are bedridden or unable to walk due to physical disabilities
* Patients with terminal cancer or human-acquired immunodeficiency syndrome
* Patients with edema (grading pitting edema +2)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2032-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of physical performance (Grip strength) | 12 weeks
  Grip strength (kg) Instrument: Smedley dynamometer
Change of physical performance(Sit to stand test) :SpO2%, HR, Borg score, times and second will be reported to present the result of Sit to stand test. | 12 weeks
  SpO2%, HR, Borg score, times and second
Change of physical performance (SPPB): Sit to stand test, balance test and 4-meter walk test will be combined to report SPPB score | 12 weeks
  Sit to stand test, balance test and 4-meter walk test will be combined to report SPPB score
Change of physical performance :6-meter walk test (second) | 12 weeks
  5. 6-miniute walk test ( SpO2%, HR, Borg score, and the walking distance will be reported to present the result of 6-miniute walk test. )
Change of physical performance :6-miniute walk test ( SpO2%, HR, Borg score, and the walking distance will be reported to present the result of 6-miniute walk test. ) | 12 weeks
  SpO2%, HR, Borg score, and the walking distance
Change of body composition: BMI(kg/m^2) | 12 weeks
Change of body composition: SMI (kg/m^2) | 12 weeks
  PBF (%), ASM (kg), LMM (kg), BMD (T-score), RASM (kg/m^2)
PBF (%) | 12 weeks
  Change of body composition
ASM (kg) | 12 weeks
  Change of body composition
LMM (kg) | 12 weeks
  Change of body composition
BMD (T-score) | 12 weeks
  Change of body composition
RASM (kg/m^2) | 12 weeks
  Change of body composition
Forced Expiratory Volume in 1 second(FEV1(L)) | 12 weeks
  Change of lung function
Forced Expiratory Volume in 1 second as a percentage of predicted value(FEV1 (%)) | 12 weeks
  Change of lung function
ratio of Forced Expiratory Volume in 1 second to Forced Vital Capacity as a percentage(FEV1/FVC (%)) | 12 weeks
  Change of lung function
Peak Expiratory Flow(PEF (L/min)) | 12 weeks
  Change of lung function
RBC (/μL) | 12 weeks
  Complete blood count
WBC (/μL) | 12 weeks
  Complete blood count
PLT (/μL) | 12 weeks
  Complete blood count
Hb | 12 weeks
  Complete blood count
Hematocrit | 12 weeks
  Complete blood count
TG | 12 weeks
  Hepatic function
SGOT (U/L) | 12 weeks
  Hepatic function
SGPT (U/L) | 12 weeks
  Hepatic function
Total cholesterol(mg/dL) | 12 weeks
  Hepatic function
LDL-C (mg/dL) | 12 weeks
  LDL-C (mg/dL)
Fasting glucose (mg/dL) | 12 weeks
  Fasting glucose (mg/dL)
HbA1c (%) | 12 weeks
  HbA1c (%)
Total protein (g/dL) | 12 weeks
  Total protein (g/dL)
Albumin (g/dL) | 12 weeks
  Albumin (g/dL)
Renal function | 12 weeks
  BUN、CREAT(mg/dL)
Hs-CRP | 12 weeks
  Hs-CRP
Vitamin D | 12 weeks
  Vitamin D

SECONDARY OUTCOMES:
SARC-Calf questionnaire | 12 weeks
  compare the effect of the same intervention on Sarcopenia and different severity of Sarcopenia.
Grip strength test | 12 weeks
  compare the outcome of physical performance of the same intervention on Sarcopenia and different severity of Sarcopenia.
Sit-stand test | 12 weeks
  compare the outcome of physical performance of the same intervention on Sarcopenia and different severity of Sarcopenia.
Short physical performance battery (SPPB) | 12 weeks
  compare the outcome of physical performance of the same intervention on Sarcopenia and different severity of Sarcopenia.
Gait speed test | 12 weeks
  compare the outcome of physical performance of the same intervention on Sarcopenia and different severity of Sarcopenia.
Six-minute walk test. | 12 weeks
  compare the outcome of physical performance of the same intervention on Sarcopenia and different severity of Sarcopenia.
Bioelectrical impedance analysis (BIA) | 12 weeks
  compare the effect of the same intervention on Sarcopenia and different severity of Sarcopenia on the outcome of body composition
SMI (kg/m^2) | 12 weeks
  DXA is an X-ray machine that can generate two types of low-energy X-rays. X-rays of different energies are attenuated to different degrees by different media. The higher the density of the medium, the greater the attenuation caused by X-rays. Through computer calculations, DXA can not only measure bone density but also analyze body composition, determining the quantity and ratio of muscle and fat. Bone density: L-spine (g/cm^2) and T-score , Femoral neck (g/cm^2) and T-score
Forced Expiratory Volume in 1 second (FEV1) | 12 weeks
  Pulmonary function
Forced Expiratory Volume in 1 second as a percentage of predicted value (FEV1 (%)) | 12 weeks
  Pulmonary function
ratio of Forced Expiratory Volume in 1 second to Forced Vital Capacity as a percentage (FEV1/FVC (%)) | 12 weeks
  Pulmonary function
Peak Expiratory Flow (PEF (L/min)) | 12 weeks
  Pulmonary function

CONTACTS AND LOCATIONS:
Overall Officials: Pin-Kuei Fu, Principal Investigator — Department of Chest Medicine of Taichung Veterans General
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan